CLINICAL TRIAL: NCT07141680
Title: Clinical and Radiographic Evaluation of Intentional Replantation Treatment in Periodontally Hopeless Teeth, Randomized Controlled Clinical Study
Brief Title: Comparison of Replantation and Splinting Alone in Lower Anterior Teeth
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Saglik Bilimleri Universitesi (Other)
Responsible Party: Principal Investigator, Tuğçe Paksoy, associate professor, Saglik Bilimleri Universitesi
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 24-7
Record Dates: First submitted 2025-08-18; First posted 2025-08-26 (Actual); Last update posted 2025-08-26 (Actual); Status verified 2025-08

CONDITIONS: Periodontitis
Keywords: intentional replantation; periodontal splint; tooth mobility; tooth reimplantation; tooth replantation
MeSH Terms: conditions — Periodontitis; Tooth Mobility | interventions — Replantation; Splints

STUDY DESIGN:
Intervention Model Description: Fifty individuals aged 18-65 with severe clinical periodontal attachment loss (>3 mm) and alveolar bone loss (⅔ or more of the root) in the anterior incisors will participate in the study, taking into account the inclusion and exclusion criteria. All patients will undergo non-surgical periodontal treatment before being divided into groups. Patients who meet the inclusion criteria for the study will be randomly selected into the experimental and control groups: 1. Control group (n=25): The group that will undergo conventional root canal treatment and be followed up with a splint. 2. Experimental group (n=25): The group that will undergo conventional root canal treatment followed by planned replantation treatment and be followed up with a splint.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Replantation (Active Comparator): Replantation group (n=25): Group that underwent conventional canal treatment followed by planned replantation treatment and splinting.
  Interventions: Procedure: Replantation
- Splint (Placebo Comparator): Splint group (n=25): The group that will undergo conventional canal treatment and splinting.
  Interventions: Procedure: Splint

INTERVENTIONS:
Procedure: Replantation — Root canal treatment Tooth extraction and replacement Splinting
  Arms: Replantation
Procedure: Splint — Root canal treatment Splinting
  Arms: Splint

SUMMARY:
Replantation is defined as the intentional extraction and repositioning of teeth that have lost their periodontal support. The aim of this study is to evaluate the clinical and radiographic follow-up results of planned replantation treatment in cases with advanced periodontal destruction and to compare it with splinting alone.

Twenty-five patients with periodontal damage in the control group and 25 patients in the experimental group will be included in the study. The clinical parameters of both groups will be evaluated at baseline, 1, 3, and 6 months using periodontal indices and the Visual Analog Scale (VAS).

DETAILED DESCRIPTION:
Fifty individuals aged 18-65 with severe clinical attachment loss (>3 mm) and alveolar bone loss (⅔ or more of the root) in their lower anterior incisors will participate in the study, taking into account the inclusion and exclusion criteria. All patients will undergo non-surgical periodontal treatment before being divided into groups. Patients who meet the inclusion criteria will be randomly selected for the experimental and control groups:

Control group (n=25): The group that will undergo conventional root canal treatment and be followed up with a splint Experimental group (n=25): The group that will undergo conventional root canal treatment followed by planned replantation treatment and splinting.

Infiltrative anesthesia is applied to the tooth planned for replantation. The tooth is extracted with care not to cause trauma to the surrounding tissues. Care is taken not to touch the root surface of the extracted tooth, especially in areas where it comes into contact with the bone apically, in order not to damage the cells that promote healing. If there are attachments on the root surface, they are removed with ultrasound. The tooth is placed in the prepared tetracycline solution and left for 5 minutes. During this time, the extraction socket is gently checked to ensure it is clean. Any granulation tissue that would prevent the tooth root from settling into the bone and making contact is removed. The tooth is removed from the tetracycline solution and placed in the socket. The tooth is stabilized and a temporary splint is applied. Contacts are removed during closure and intrusive movements. The patient is informed that they should not bite or tear with their front teeth and that they should protect the tooth. After 2 weeks, a permanent periodontal splint will be applied.

The clinical parameters of the patients participating in the study will be monitored for 6 months, and the success of the planned replantation treatment will be evaluated by comparing the data from the control group and the test group. It will be investigated whether there is a significant difference between the treatments applied to the control and test groups in terms of clinical and radiographic findings and patient satisfaction.

ELIGIBILITY:
Inclusion Criteria:

* All patients are systemically healthy or have their systemic conditions under control.
* Lower anterior incisors (42, 41, 31, 32) will be included.
* Mobility classification will be Miller 3.
* Radiograph showing 50% or more bone loss at the root.
* Probing depth of 5 mm or more.
* Bone level of adjacent teeth at ⅔ or better than the root.
* Mobility of adjacent teeth will be Miller 0 or Miller 1.
* The patient prefers to keep the tooth in the mouth rather than having it extracted.

Exclusion Criteria:

* Systemic Comorbidity
* Smoking
* Root Resorption
* Root Fracture or Crack
* Ankylosis of the Tooth

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-05-24 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Clinical attachment loss (CAL) | Baseline, 3rd and 6th months
  CAL is measured as the change in distance from the cementoenamel junction to the bottom of the gingival sulcus (the most coronal attachment) using a Williams periodontal probe. The changes in clinical attachment loss was measured for determining the severity of disease.
Bone Loss,(BL) | Baseline and 6th monts
  The pre- and post-treatment tooth length/bone ratio around the tooth root will be determined using CBCT and periapical radiographs. The amount of bone loss (% bone loss, BL) will be determined using a millimeter scale from both the mesial and distal regions of the teeth, according to the method described by Schulte and colleagues (10) using periapical radiographs. To determine individual bone loss, intra-alveolar root length (hi) and total root length (hg) are measured. Hg, the total root length, is defined as the distance from the apex to the proximal enamel-cementum junction, parallel to the long axis of the teeth. Since the distance between the alveolar bone crest and the enamel-cementum junction varies between 0.75 and 1.49 mm, 1.5 mm is subtracted from the total root length during calculation. The intra-alveolar root length is defined as the distance from the apex to the highest point on the alveolar margin. The change in bone loss at baseline and at 6 months will be examined.

SECONDARY OUTCOMES:
Probing pocket depth (PPD) | Baseline, 3rd and 6th months
  Probing pocket depth (PPD) measured as the change in distance from the gingival margin to the bottom of the gingival sulcus using a Williams periodontal probe.
Bleeding on probing (BOP) | Baseline, 3rd and 6th months
  All six sites of all teeth were probed to assess whether this elicited bleeding (+) or not (-). The severity of gingival inflammation was expressed as a percentage (BOP=number of bleeding sites×100/number of sites evaluated).
Mobility | Baseline, 3rd and 6th months
  Tooth mobility will be assessed using a 5N (500g) manual measurement. Changes in mobility will be examined with treatment.
  0th degree: no mobility
  1. st degree: slight movement
  2. nd degree: up to 1 mm
  3. rd degree: more than 1 mm and movement in all directions vertical mobility
Gingival index (GI) | Baseline, 3rd and 6th months
  To determine the gingival index (Löe & Silness), gingival bleeding caused by running a Williams periodontal probe inside the pocket on the mesial, distal, buccal, and palatal surfaces of all teeth was evaluated. The gingival index of an individual was obtained by summing the values determined for each tooth and calculating the averages. Scoring was as follows:
  0: Healthy gums.
  1. Mild discolouration and oedematous gingiva. No bleeding on probing.
  2. Red, oedematous and shiny gingiva. There is bleeding on probing.
  3. Red, oedematous and ulcerated gingiva. There is spontaneous bleeding. Gingival index was recorded for classifying and evaluating sulcular gingival inflammation.
Plaque index (PI) | Baseline, 3rd and 6th months
  Patients' plaque indices will be recorded according to the Silness and Löe plaque index. After the teeth are dried with air, the amount of plaque near the gingival margin of each tooth is examined with an inspection and examination probe. Index values between 0 and 3 are given according to the amount of plaque on the tooth surface.
  According to this index:
  0: No plaque.
  1. A thin layer of plaque is observed along the gingival margin. This thin layer can be detected with an examination probe.
  2. A moderate layer of plaque is observed along the gingival margin. The plaque in question can be detected with the naked eye.
  3. A significant amount of plaque is observed along the gingival margin, and the interdental spaces are filled with plaque.
VAS measurement values | Baseline, 3rd and 6th months
  VAS is the most commonly used scale for measuring pain intensity and tracking the degree of pain relief. VAS is a 10 cm line with the extremes of "no pain" and "worst possible pain," and the measurement is determined by the patient marking the line that best describes their pain intensity. The average of the values obtained for patients is calculated.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Health Sciences, Hamidiye Faculty of Dentistry., Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
There is no need for such a sharing